CLINICAL TRIAL: NCT00772941
Title: Drug Use Investigation Of Champix (Regulatory Post Marketing Commitment Plan)
Brief Title: Drug Use Investigation Of Varenicline (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3051109
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Varenicline: Patients taking Varenicline.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Champix Tablets 0.5mg or Champix Tablets 1mg, depending on the Investigator prescription.
  Frequency and duration are according to Package Insert as follows.
  "The usual adult dosage for oral use is 0.5 mg of varenicline once daily after eating for days 1 to 3, 0.5 mg twice daily after eating in the morning and evening for days 4 to 7, and 1 mg twice daily after eating in the morning and evening on and after day 8. The drug should be administered to patients for 12 weeks."
  Other Names: Champix, Chantix

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Varenicline(Champix) should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Varenicline(Champix) in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Varenicline(Champix).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A3051109 prescribes the Varenicline(Champix).
Sampling Method: Probability Sample
Enrollment: 3939 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051109&StudyName=Drug%20Use%20Investigation%20Of%20Varenicline%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Participants taking Varenicline according to Japanese Package Insert.
Period: Overall Study
Arm/Group | Varenicline
Started | 3939
Completed | 3257
Not Completed | 682
Not completed — CRFs not available | 195
Not completed — Study not completed | 16
Not completed — Missed Visits | 374
Not completed — Poor Compliance | 7
Not completed — GPSP Violation | 90

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 3257
Age, Customized [Number; unit: Participants]
  <65 years | 2768
  >=65 years | 489
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1078
  Male | 2179

OUTCOME MEASURES:

1. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events - Gender.
Description: Number of participants with Treatment Related Adverse Events of Varenicline to determine whether gender is a significant risk factor.
Time Frame: 24 weeks
Population: The safety analysis population consists of the participants who satisfy the case conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Groups:
- Male: Male participants taking Varenicline according to Japanese Package Insert.
- Female: Female participants taking Varenicline according to Japanese Package Insert.
Arm/Group | Male | Female
Number analyzed (Participants) | 2179 | 1078
participants | 377 | 336
Statistical Analysis 1: Comparison: Male vs Female; The risk factor tested was "Gender". The null hypothesis is that there is no difference between "Male and Female" in the frequency of Treatment Related Adverse Events; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events - Age.
Description: Number of participants with Treatment Related Adverse Events of Varenicline to determine whether age is a significant risk factor.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- <65 Years: Participants with <65 years taking Varenicline according to Japanese Package Insert.
- >=65 Years: Participants with >=65 years taking Varenicline according to Japanese Package Insert.
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 2768 | 489
participants | 571 | 142
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; The risk factor tested was "Age". The null hypothesis is that there is no difference between "<65 years and >=65 years" in the frequency of Treatment Related Adverse Events; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events - Chronic Obstructive Pulmonary Disease as a Complication.
Description: Number of participants with Treatment Related Adverse Events of Varenicline to determine whether Chronic obstructive pulmonary disease as a complication is a significant risk factor.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Varenicline - With Chronic Obstructive Pulmonary Disease: Participants with chronic obstructive pulmonary disease as a complication taking Varenicline according to Japanese Package Insert.
- Varenicline - Without Chronic Obstructive Pulmonary Disease: Participants without chronic obstructive pulmonary disease as a complication taking Varenicline according to Japanese Package Insert.
Arm/Group | Varenicline - With Chronic Obstructive Pulmonary Disease | Varenicline - Without Chronic Obstructive Pulmonary Disease
Number analyzed (Participants) | 46 | 3211
participants | 23 | 690
Statistical Analysis 1: Comparison: Varenicline - With Chronic Obstructive Pulmonary Disease vs Varenicline - Without Chronic Obstructive Pulmonary Disease; The risk factor tested was "Chronic obstructive pulmonary disease as a complication". The null hypothesis is that there is no difference between "Varenicline with and without Chronic obstructive pulmonary disease as a complication" in the frequency of Treatment Related Adverse Events; Test type: Superiority or Other; p < 0.001, Chi-squared

4. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events - Concomitant Drugs.
Description: Number of participants with Treatment Related Adverse Events of Varenicline to determine whether taking concomitant drugs is a significant risk factor.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Varenicline - With Concomitant Drugs: Participants taking concomitant drugs while taking Varenicline according to Japanese Package Insert.
- Varenicline - Without Concomitant Drugs: Participants taking no concomitant drugs while taking Varenicline according to Japanese Package Insert.
Arm/Group | Varenicline - With Concomitant Drugs | Varenicline - Without Concomitant Drugs
Number analyzed (Participants) | 738 | 2519
participants | 289 | 424
Statistical Analysis 1: Comparison: Varenicline - With Concomitant Drugs vs Varenicline - Without Concomitant Drugs; The risk factor tested was "concomitant drugs". The null hypothesis is that there is no difference between "Varenicline with and without concomitant drugs" in the frequency of Treatment Related Adverse Events; Test type: Superiority or Other; p < 0.001, Chi-squared

5. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events - Concomitant Therapies.
Description: Number of participants with Treatment Related Adverse Events of Varenicline to determine whether receiving concomitant therapies is a significant risk factor.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Varenicline - With Concomitant Therapies: Participants receiving concomitant therapies while taking Varenicline according to Japanese Package Insert.
- Varenicline - Without Concomitant Therapies: Participants receiving no concomitant therapies while taking Varenicline according to Japanese Package Insert.
Arm/Group | Varenicline - With Concomitant Therapies | Varenicline - Without Concomitant Therapies
Number analyzed (Participants) | 101 | 3156
participants | 45 | 668
Statistical Analysis 1: Comparison: Varenicline - With Concomitant Therapies vs Varenicline - Without Concomitant Therapies; The risk factor tested was "concomitant therapies". The null hypothesis is that there is no difference between "Varenicline with and without concomitant therapies" in the frequency of Treatment Related Adverse Events; Test type: Superiority or Other; p < 0.001, Chi-squared

6. Primary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events - Weight at Baseline.
Description: Number of participants with Treatment Related Adverse Events to determine whether weight at baseline is a significant risk factor.
Time Frame: 24 weeks
Population: The safety analysis population consists of the participants who satisfy the case conditions and in whom administration of this drug was confirmed. The number of participants who provided weight data at baseline was 1700.
Measure: Number; unit: participants
Groups:
- <40 kg at Baseline: Participants whose weights at baseline were less than 40 kg.
- >=40 kg and <50 kg at Baseline: Participants whose weights at baseline were more than or equal to 40 kg and less than 50 kg.
- >=50 kg and <60 kg at Baseline: Participants whose weights at baseline were more than or equal to 50 kg and less than 60 kg.
- >=60 kg and <70 kg at Baseline: Participants whose weights at baseline were more than or equal to 60 kg and less than 70 kg.
- >=70 kg and <80 kg at Baseline: Participants whose weights at baseline were more than or equal to 70 kg and less than 80 kg.
- >= 80 kg at Baseline: Participants whose weights at baseline were more than or equal to 80 kg.
Arm/Group | <40 kg at Baseline | >=40 kg and <50 kg at Baseline | >=50 kg and <60 kg at Baseline | >=60 kg and <70 kg at Baseline | >=70 kg and <80 kg at Baseline | >= 80 kg at Baseline
Number analyzed (Participants) | 13 | 215 | 453 | 497 | 342 | 180
participants | 6 | 98 | 135 | 110 | 61 | 31
Statistical Analysis 1: Comparison: <40 kg at Baseline vs >=40 kg and <50 kg at Baseline vs >=50 kg and <60 kg at Baseline vs >=60 kg and <70 kg at Baseline vs >=70 kg and <80 kg at Baseline vs >= 80 kg at Baseline; The risk factor tested was "Weight at Baseline". The null hypothesis is that there is no association between "Weight at Baseline and the frequency of Treatment Related Adverse Events"; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: <40 kg at Baseline vs >=40 kg and <50 kg at Baseline vs >=50 kg and <60 kg at Baseline vs >=60 kg and <70 kg at Baseline vs >=70 kg and <80 kg at Baseline vs >= 80 kg at Baseline; The risk factor tested was "Weight at Baseline". The null hypothesis is that there is no linear trend in the frequency of Treatment Related Adverse Events across increasing levels of Weight at Baseline; Test type: Superiority or Other; p < 0.001, Cochran-Armitage

7. Primary Outcome: Risk Factors for the Proportion of Responders - Tobacco Consumption Per Day.
Description: The primary analysis item was "the number of participants succeeding with continuous smoking cessation for the previous 4 weeks/the number of participants for efficacy evaluation excluding drop-out participants.
Time Frame: 24 weeks
Population: The efficacy analysis population basically consists of the evaluable participants in accordance with the separately prepared analysis plan (participants judged to have been evaluated appropriately). The number of participants who provided data on daily tobacco consumption was 2827.
Measure: Number; unit: participants
Groups:
- <=20 Cigarettes Per Day: Participants with <=20 cigarettes per day during treatment with Varenicline according to Japanese Package Insert.
- >=21 and <=40 Cigarettes Per Day: Participants with >=21 and <=40 cigarettes per day during treatment with Varenicline according to Japanese Package Insert.
- >=41 Cigarettes Per Day: Participants with >=41 cigarettes per day during treatment with Varenicline according to Japanese Package Insert.
Arm/Group | <=20 Cigarettes Per Day | >=21 and <=40 Cigarettes Per Day | >=41 Cigarettes Per Day
Number analyzed (Participants) | 1637 | 1082 | 108
participants | 1299 | 817 | 66
Statistical Analysis 1: Comparison: <=20 Cigarettes Per Day vs >=21 and <=40 Cigarettes Per Day vs >=41 Cigarettes Per Day; The risk factor tested was "Tobacco consumption per day". The null hypothesis is that there is no association between "Tobacco consumption per day and the efficacy of Varenicline"; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: <=20 Cigarettes Per Day vs >=21 and <=40 Cigarettes Per Day vs >=41 Cigarettes Per Day; The risk factor tested was "Tobacco consumption per day". The null hypothesis is that there is no linear trend in the efficacy of Varenicline across increasing levels of tobacco consumption per day; Test type: Superiority or Other; p < 0.001, Cochran-Armitage

8. Primary Outcome: Risk Factors for the Proportion of Responders - Prolonged Administration After 12 Weeks.
Description: as for outcome 7
Time Frame: 24 weeks
Population: The efficacy analysis population basically consists of the evaluable participants in accordance with the separately prepared analysis plan (participants judged to have been evaluated appropriately). The number of participants in whom the prolonged administration of Varenicline after 12 weeks was confirmed was 2598.
Measure: Number; unit: participants
Groups:
- Administration Prolonged After 12 Weeks: Participants with prolonged administration of Varenicline after 12 weeks according to Japanese Package Insert.
- Administration Not Prolonged After 12 Weeks: Participants without prolonged administration of Varenicline after 12 weeks according to Japanese Package Insert.
Arm/Group | Administration Prolonged After 12 Weeks | Administration Not Prolonged After 12 Weeks
Number analyzed (Participants) | 64 | 2534
participants | 39 | 1993
Statistical Analysis 1: Comparison: Administration Prolonged After 12 Weeks vs Administration Not Prolonged After 12 Weeks; The risk factor tested was "prolonged administration after 12 weeks". The null hypothesis is that there is no difference between "administration prolonged after 12 weeks and administration not prolonged after 12 weeks" in the efficacy of Varenicline; Test type: Superiority or Other; p < 0.001, Chi-squared

9. Primary Outcome: Risk Factors for the Proportion of Responders - Antipsychotics as a Concomitant Drug.
Description: as for outcome 7
Time Frame: 24 weeks
Population: The efficacy analysis population basically consists of the evaluable participants in accordance with the separately prepared analysis plan (participants judged to have been evaluated appropriately). The number of participants who provided data on concomitant administration of antipsychotics was 2842.
Measure: Number; unit: participants
Groups:
- Varenicline - With Antipsychotics as a Concomitant Drug: Varenicline with Antipsychotics as a Concomitant Drug
- Varenicline - Without Antipsychotics as a Concomitant Drug: Varenicline without Antipsychotics as a Concomitant Drug
Arm/Group | Varenicline - With Antipsychotics as a Concomitant Drug | Varenicline - Without Antipsychotics as a Concomitant Drug
Number analyzed (Participants) | 140 | 2702
participants | 85 | 2111
Statistical Analysis 1: Comparison: Varenicline - With Antipsychotics as a Concomitant Drug vs Varenicline - Without Antipsychotics as a Concomitant Drug; The risk factor tested was "antipsychotics as a concomitant drug". The null hypothesis is that there is no difference between "Varenicline with and without antipsychotics as a concomitant drug" in the efficacy of Varenicline; Test type: Superiority or Other; p < 0.001, Chi-squared

10. Primary Outcome: Number of Participants With Treatment Related Adverse Events.
Description: Adverse events mean all unfavorable events that occur in participants after administration of Varenicline, irrespective of causal relationship to Varenicline (including clinically problematic abnormal changes in laboratory test values). Treatment related Adverse Events were evaluated in company with the causal relationship to Varenicline. The safety was evaluated on the first visit after 24 weeks; however, it was evaluated on the last visit for those who had stopped visiting before 24 weeks.
Time Frame: 24 weeks
Population: No statistical analysis provided for the frequency of treatment related adverse events.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 3257
participants | 713

11. Primary Outcome: Number of Unlisted Treatment Related Adverse Events According to Japanese Package Insert.
Description: Adverse events mean all unfavorable events that occur in participants after administration of Varenicline, irrespective of causal relationship to Varenicline (including clinically problematic abnormal changes in laboratory test values). Numbers of Treatment Related Adverse Events were evaluated in company with the causal relationship to Varenicline. Unlisted treatment related adverse events were confirmed with listed adverse drug reaction in Japanese package insert. The safety was evaluated on the first visit after 24 weeks; however, it was evaluated on the last visit for those who had stopped visiting before 24 weeks.
Time Frame: 24 weeks
Population: No statistical analysis provided for the frequency of unlisted treatment related adverse events.
Measure: Number; unit: events
Arm/Group | Varenicline
Number analyzed (Participants) | 3257
events | 30

12. Secondary Outcome: Number of Participants With Continuous Abstinence Situation by 52 Weeks.
Description: Number of participants with dependence on Varenicline by 52 weeks. Varenicline-dependent Treatment Related Adverse Events are Feeling abnormal, Feeling drunk, Feeling jittery, Disturbance in attention, Dizziness, Memory impairment, Mental impairment, Psychomotor hyperactivity, Sedation, Somnolence, Confusional state, Depersonalisation, Disorientation, Dissociation, Euphoric mood, Mood variable, Mood swings, and Hallucination.
Time Frame: 52 weeks
Population: No statistical analysis provided for the frequency of Varenicline-dependent treatment related adverse events.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 3257
participants | 38

ADVERSE EVENTS:
Description: The frequency of treatment related adverse events during the study.
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 8/3257
Other Adverse Events (participants affected / at risk) | 708/3257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=3257)
Depression (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=3257)
Herpes virus infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Oral herpes (Infections and infestations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Depression (Psychiatric disorders) | 6 (6)
Nightmare (Psychiatric disorders) | 8 (8)
Abnormal dreams (Psychiatric disorders) | 9 (9)
Decreased activity (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Social avoidant behaviour (Psychiatric disorders) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1)
Bulimia nervosa (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 3 (3)
Terminal insomnia (Psychiatric disorders) | 1 (1)
Middle insomnia (Psychiatric disorders) | 1 (1)
Anger (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 2 (2)
Dysphoria (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 51 (51)
Apathy (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 3 (3)
Depressive symptom (Psychiatric disorders) | 6 (6)
Restlessness (Psychiatric disorders) | 1 (1)
Somnolence (Nervous system disorders) | 23 (23)
Headache (Nervous system disorders) | 35 (35)
Dementia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 13 (13)
Migraine (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Peripheral coldness (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 397 (397)
Gastritis (Gastrointestinal disorders) | 49 (49)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 10 (10)
Flatulence (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 22 (22)
Glossitis (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 18 (18)
Abdominal distension (Gastrointestinal disorders) | 12 (12)
Constipation (Gastrointestinal disorders) | 91 (91)
Vomiting (Gastrointestinal disorders) | 39 (39)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2)
Lactation disorder (Reproductive system and breast disorders) | 1 (1)
Irritability (General disorders) | 6 (6)
Feeling abnormal (General disorders) | 3 (3)
Chest discomfort (General disorders) | 1 (1)
Malaise (General disorders) | 10 (10)
Thirst (General disorders) | 4 (4)
Pyrexia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Blood pressure increased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Weight increased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.